CLINICAL TRIAL: NCT03242213
Title: Patient Management of Depression Through Technology: a Study of Digitally Enabled Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AHC6680
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Standard of Care
- Mobile App (Active Comparator): Standard of Care and Mobile App
  Interventions: Behavioral: Mobile App

INTERVENTIONS:
Behavioral: Mobile App — The intervention in this study is a mobile health app, which provides patients with a way to track emotional wellbeing and depression symptoms, set up medication reminders, track adherence to medications, record side effects experienced, and take surveys/tests to assess cognitive symptoms and depression.
  Arms: Mobile App

SUMMARY:
The current randomized controlled trial is a pilot study that will assess the effectiveness and feasibility of a mobile phone application intervention. The objective is to determine whether the use of a mobile health application for patient self-management of depression improves patient-provider engagement for patients diagnosed with major depressive disorder.

DETAILED DESCRIPTION:
This pilot study will be a randomized, real-world effectiveness study. Patients diagnosed with major depressive disorder starting a new prescription for an antidepressant monotherapy will be eligible for participation. The study will enroll 40 patients (20 in an observational arm of usual care and 20 with access to a mobile health application). No intervention will occur in the usual care arm. The intervention in this study is a mobile health app, which provides patients with a way to track emotional wellbeing and depression symptoms, set up medication reminders, track adherence to medications, record side effects experienced, and take surveys/tests to assess cognitive symptoms and depression. Patient reported outcomes and clinical data will be collected at baseline and at study primary endpoint (18 weeks) to assess changes over time and between groups for: patient-provider engagement, disease severity, quality of life, employment productivity, cognitive function, resource utilization, and medication adherence. Additionally, resource utilization will be assessed at the one year time point. A Student's t test, if allowed for by the data distribution, will be used to assess between group differences in patient reported outcome scales assessing patient-provider engagement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70
* Ability to consent and participate in study (technical requirements for app: iPhone version 5 or later, active data plan or regular WiFi access)
* Diagnosis with major depressive disorder
* PHQ-9 score greater than 5 at baseline
* Recent (0-14 days) start on monotherapy depression medication (either new prescription or a change from a previous medication)
* Outpatient care provided by participating Advocate Medical Group clinics

Exclusion Criteria:

* Diagnosis with major psychiatric disorder (e.g. bipolar disorder, manic depressive disorder)
* Contraindications to use of depression medications
* Patients with treatment resistant depression [defined as patients who have not responded to two or more separate different antidepressant monotherapy trials of adequate dose and duration (6 weeks or longer) in the current depressive episode]
* Considered at imminent risk for hospitalization due to severe depression in the opinion of the treating physician
* History of hospitalization due to major depressive disorder in prior 3 months
* Significant risk of suicide according to the treating physician's clinical judgment or previous suicide attempt in prior 6 months
* History of response only to combination or augmentation therapy in current depressive episode
* Receipt of any investigational compound in prior 30 days (or five half-lives, whichever is longer)
* Current participation in another clinical study
* Lack of functional English literacy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Patient activation | 18 weeks
  This will be assessed by the Patient Activation Measure, a validated scale that measures patient knowledge, skills and confidence in disease self-management in the primary care setting.
Patient-provider engagement | 18 weeks
  This will be assessed by the Patient-Provider Engagement Scale (PPES-7), an instrument developed for this study to measure patient knowledge, communication, and interaction with their provider specific to depression management.

SECONDARY OUTCOMES:
Depression symptoms | 18 weeks
  This patient reported outcome is assessed by the clinical depression severity. PHQ-9 scale, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Cognitive dysfunction | 18 weeks
  This patient reported outcome is assessed by the cognitive dysfunction PDQ-D scale.
Medication changes | 18 weeks
  This outcome will be assessed by clinical data on the frequency and types of medication switches.
WHO-5 survey | 18 weeks
  This patient reported outcome is assessed by the quality of life WHO-5 survey.
Health care utilization | 18 weeks
  This patient reported outcome is assessed by the healthcare resource utilization and cost RUQ-D survey.

OTHER OUTCOMES:
Long-term follow health care utilization | 1 year
  This patient reported outcome is assessed by the healthcare resource utilization and cost RUQ-D survey.

CONTACTS AND LOCATIONS:
Overall Officials: David Kemp, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCue M, Blair C, Fehnert B, King J, Cormack F, Sarkey S, Eramo A, Kabir C, Khatib R, Kemp D. Mobile App to Enhance Patient Activation and Patient-Provider Communication in Major Depressive Disorder Management: Collaborative, Randomized Controlled Pilot Study. JMIR Form Res. 2022 Oct 27;6(10):e34923. doi: 10.2196/34923. PMID 36301599